CLINICAL TRIAL: NCT07186413
Title: A Multicenter, Randomized, Double-blinded, Parallel-group, Vehicle-controlled Study to Compare the Efficacy, Safety and Pharmacokinetics of Trifarotene 50 mcg/g Cream in Chinese Subjects With Acne Vulgaris
Brief Title: A Study to Compare the Efficacy, Safety and Pharmacokinetics of Trifarotene 50 mcg/g Cream in Chinese Subjects With Acne Vulgaris
Acronym: AKLIEF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD5789.SPR.205101
Record Dates: First submitted 2025-08-26; First posted 2025-09-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trifarotene Cream (Experimental): Participants will apply Trifarotene 50 mcg/g cream once daily (QD) in the evening for 12 weeks.
  Interventions: Drug: Trifarotene
- Vehicle Cream (Active Comparator): Participants will apply Vehicle cream QD in the evening for 12 weeks.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Trifarotene — Trifarotene cream applied QD topically.
  Other Names: CD5789
  Arms: Trifarotene Cream
Drug: Vehicle Cream — Vehicle cream applied QD topically.
  Arms: Vehicle Cream

SUMMARY:
The primary objective is to assess the efficacy of trifarotene 50 microgram per gram (mcg/g) cream versus vehicle cream when applied once daily (QD) for 12 weeks in Chinese participants with moderate facial and truncal acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria to be included in the study:

1. Male or female Chinese participants aged 9 years or older at the screening visit.
2. A minimum of 20 inflammatory lesions and 25 non-inflammatory lesions on the face at Screening and Baseline.
3. Facial acne vulgaris severity grade 3 (moderate) on the IGA scale at Screening and Baseline.
4. A minimum of 20 inflammatory lesions and 20 non-inflammatory lesions but no more than 100 non-inflammatory lesion counts on the trunk (shoulders, upper back, and upper anterior chest) reachable for self-application of investigational product by the participant at Screening and Baseline (optional criterion for participant between 9 and 11 years of age).
5. Acne vulgaris severity grade 3 (moderate) on the PGA scale at Screening and Baseline visits on trunk (shoulders, upper back and upper anterior chest) reachable for self-application of investigational product by the participant (optional criterion for participants between 9 and 11 years of age).
6. Female participants of non-childbearing potential, i.e., premenstrual, or postmenopausal. Postmenopausal participants must meet one criterion at Screening:

   * Absence of menstrual bleeding for 1 year before screening with no other medical reason, confirmed with follicle-stimulating hormone level in the postmenopausal range.
   * Documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at least 3 months before Screening.
7. Female participants of childbearing potential (i.e., fertile, after menarche and until becoming postmenopausal unless permanently sterile) must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test (UPT) at the baseline visit (with a sensitivity of 25 international units per litre [IU/L] or less). They must use at least 1 adequate and approved method of contraception throughout the study and for 1 month after the last dose of investigational product.
8. Premenstrual participants who start menses during the study must use at least 1 adequate and approved method of contraception throughout the study and for 1 month after the last dose of investigational product.
9. Willing and able to comply with all the time commitments and procedural requirements of the clinical study protocol.
10. Understands and signs an informed consent form (ICF) at the screening visit, before any investigational procedures are performed.
11. Participants who are younger than 18 years of age and whose parent/legal representative is willing/able to comply with the study requirements and understand/sign the ICF at the screening visit, before any investigational procedures are performed, will sign the assent ICF at the screening visit.
12. At selected clinical sites: If a participant who is 18 years of age or older at the screening visit and agrees to participate in study photographs, verified by dating and signing a separate approved photography ICF. For participants younger than 18 years of age, an assent photography ICF signed by the participant in conjunction with a photography ICF signed by the parents(s)/legal representative at the screening visit.
13. Participant is informed of terms pertaining to personal information protection and privacy and is willing to share personal information and data, in accordance with local regulations.

Exclusion Criteria:

Participants meeting the following criteria at the screening or baseline visits are ineligible to participate in this study:

1. Pregnant women (positive serum pregnancy test result at the screening visit or positive UPT at the baseline visit), breastfeeding women, or women planning a pregnancy during the study or within 1 month after the last investigational product application.
2. Severe forms of acne (e.g., acne conglobata, acne fulminans) or secondary acne form (e.g., chloracne, drug-induced acne) at the screening and baseline visits.
3. More than 1 nodule on the face at the screening and baseline visits.
4. More than 1 nodule on the trunk at the screening and baseline visits.
5. Any acne cyst on the face at the screening and baseline visits.
6. Any acne cyst on the trunk at the screening and baseline visits.
7. Facial or truncal hair that may interfere with the study assessments according to investigator's judgment.
8. Abnormal pigmentation, wound, scar, or tattoo on the face or on the shoulders, upper back, or chest that may interfere with the study assessments according to investigator's judgment.
9. Any uncontrolled or serious disease or any medical or surgical condition that may interfere with the interpretation of the study results and/or put the participant at significant risk according to investigator's judgment.
10. Abnormal laboratory test results at the screening visit (hematology, comprehensive metabolic panel, and urinalysis) judged as clinically significant by the investigator (to be checked before the baseline visit), which may interfere with the interpretation of the study results and/or put the participant at significant risk (e.g., elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) (> 3 × upper limit of normal [ULN])).
11. Known allergies or hypersensitivities to any component of the formulation of the investigational products (trifarotene 50 mcg/g cream or vehicle cream; see Investigator's Brochure).
12. Previously participated in any trifarotene cream clinical study.
13. Current participation in any other clinical study of a drug or device OR past participation within 30 days before the baseline visit.
14. Alcohol or drug abuse or substance dependence within 12 months before the screening visit.
15. Inability or unwillingness to undergo multiple venipunctures because of poor tolerability or venous access.
16. Loss of over 500 mL of blood or blood donation within the last 3 months before the screening visit.
17. Having received prohibited medication or treatment during the study.
18. Exposure to excessive ultraviolet (UV) radiation within 1 month before the baseline visit.
19. Unwillingness to avoid excessive or prolonged exposure to UV light (i.e., occupational exposure to the sun, sunbathing, tanning bed use, phototherapy) throughout the study.
20. Any drug that in the opinion of the investigator may interfere with the study assessments or exacerbate acne, i.e., lithium, halogens, haloperidol, hydantoin, phenobarbital, Vitamin B12, androgens.
21. Unwillingness to refrain from prohibited medication during the clinical study as defined by protocol.
22. Participant vulnerability (such as freedom deprivation, mental disease, those incapable of giving consent) as defined in Section 1.61 of the International Council for Harmonization Guideline for Good Clinical Practice (GCP).
23. More than 1 participant sharing the same household.
24. Clinical site personnel, close relatives of the clinical site personnel (e.g., parents, children, siblings, or spouse), employees, or close relatives of employees of the Sponsor company.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 561 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Investigator Global Assessment (IGA) Success (Face only) at Week 12 | Baseline to Week 12
  The areas defined for IGA assessment are the forehead, each cheek, chin, and nose. IGA will be confined to a global assessment of each area defined above. IGA consists of 5 grades ranging from 0-4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Success Rate, defined as the percentage of participants who achieve an IGA score (face only) of 1 (Almost Clear) or 0 (Clear) and at least a 2-grade improvement from Baseline to Week 12.
Change from Baseline to Week 12 in Facial Non-inflammatory Lesion Count | Baseline to Week 12
Change from Baseline to Week 12 in Facial Inflammatory Lesion Count | Baseline to Week 12

SECONDARY OUTCOMES:
Percentage of Participants with Physician Global Assessment (PGA) Success at Week 12 | Baseline to Week 12
  The areas defined for PGA assessment are shoulders, upper back and upper anterior chest which are accessible to self-application by the participants. PGA will be confined to a global assessment of each areas defined above. The PGA is a snapshot static assessment to be done prior to detailed lesion counts. PGA consists of 5 grades ranging from 0-4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. PGA Success, defined as the percentage of participants who achieve a PGA score of 1 (Almost Clear) or 0 (Clear) and at least a 2-grade improvement from Baseline to Week 12
Change from Baseline to Week 12 in Truncal Non-inflammatory Lesion Count | Baseline to Week 12
Change from Baseline to Week 12 in Truncal Inflammatory Lesion Count | Baseline to Week 12
Number of Participants With Adverse Events (AEs), Including AEs of Special Interest (AESIs), Treatment-emergent AEs (TEAEs), and Serious AEs (SAEs) | Baseline to Week 12
Investigator's Local Tolerability Assessment | Baseline, Weeks 1, 2, 4, 8 and 12
  Local tolerability, which includes individual assessment of erythema, scaling, dryness, and stinging/burning, will be graded on a 4-point scale (ranging from 0 [None] to 3 [Severe]) separately for the face and trunk. A higher score indicated a severe outcome. The areas for evaluation on the face include the forehead, nose, chin, and right and left cheeks. The areas for evaluation on the upper trunk include the shoulders, right and left chest, and right and left upper back, which are accessible to self-application by the subject. If IP is applied to the middle and/or lower back, the local tolerability assessment of the trunk will include the upper, middle, and/or lower back, if applicable, and will be analyzed as 1 area.
Observed Plasma Concentration (Ct) in Selected Participants | Baseline, Week 4 and Week 12
  Three PK samples will be collected to inform trifarotene exposure in adult participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Galderma Research & Development Site #5378, Shanghai, Jing'an District, China

IPD SHARING:
Plan to Share IPD: Undecided